CLINICAL TRIAL: NCT05376501
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Supplemental Astaxanthin in Healthy Female Adult Participants
Brief Title: A Study to Evaluate the Effect of Astaxanthin in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: L01-21-01-T0022
Record Dates: First submitted 2022-05-10; First posted 2022-05-17 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Inflammation; Antioxidant Effect; C-Reactive Protein; Skin; Oxidative Stress; Cholesterol; Aging
MeSH Terms: conditions — Inflammation | interventions — astaxanthine

STUDY DESIGN:
Intervention Model Description: Randomization at 1:1 ratio for active or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Experimental): Active Ingredient:
  Astaxanthin
  Inactive ingredients:
  Modified food starch, sucrose, water, sodium ascorbate, DL- alpha tocopherols
  Interventions: Dietary Supplement: Astaxanthin
- Placebo (Placebo Comparator): Modified food starch, sucrose, hylocereus polyrhizus (pitaya) concentration
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin — 8 mg Astaxanthin per capsule, taken once a day with meal
  Arms: Astaxanthin
Other: Placebo — Modified food starch
  Arms: Placebo

SUMMARY:
Astaxanthin is recognized as a bioactive compound with potential benefits for human health. This study aims to evaluate a specific nutritional supplement impact on markers of oxidative stress, inflammation, lipid levels, blood flow, visual skin markers, measures of longevity, mood and skin condition.

DETAILED DESCRIPTION:
A healthy diet is characterized by a high intake of various bioactive compounds usually found in natural, organic, and fresh foodstuffs. Among these bioactive compounds, astaxanthin, a red carotenoid pigment especially found in seafood, has been recognized in the scientific literature as a potential nutraceutical due to its antioxidant, anti-inflammatory, and neurotrophic properties. Previous studies have demonstrated reduced markers of oxidative stress and inflammation and improved blood rheology. Additionally, astaxanthin help maintain healthy skin.

This randomized, double-blind, placebo-controlled study will evaluate the impact of Astaxanthin supplemented for 12 weeks, on oxidative stress, inflammation, lipid levels, blood flow, skin hydration, visual skin markers, measures of longevity, mood states and facial skin satisfaction in healthy female adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female adult participants who are 18 to 50 years of age (inclusive)
2. Have a body mass index between 18.0 to 34.9 kg/m2 (inclusive)
3. In good general health (no active or uncontrolled diseases or conditions)
4. Participants must have negative urine pregnancy test result at baseline and agree to use acceptable birth control methods during the study
5. Willing to refrain from changing their diet or lifestyle significantly for the duration of the study.
6. Agree to refrain from treatments in the defined timeframe, as outlined in the protocol
7. Willing and able to agree to the requirements and restrictions of this study, willing to give voluntary consent, able to understand and read the questionnaires, carry out all study related procedures, communicate effectively with the study staff, and agree to allow all study related evaluations

Exclusion Criteria:

1. Females who are lactating, pregnant or planning to become pregnant during the study duration
2. Have a known allergy or hypersensitivity to astaxanthin or related carotenoids, including canthaxanthin, or have hypersensitivity to an astaxanthin source, such as Haematococcus pluvialis and known sensitivity, intolerability, or allergy to any of the study products or their excipients
3. Received a vaccine for COVID-19 in the 2 weeks prior to screening, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (i.e., individuals with a history of probable or confirmed SARSCoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis)
4. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study
5. Participants with positive medical history of heart disease/cardiovascular disease, kidney disease, hepatic impairment or disease, or any other medical condition or diagnosis that the investigator would deem exclusionary
6. Participant with a positive medical history of unstable thyroid disease, immune disorder (i.e., HIV/AIDS), osteoporosis, a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit)
7. Participants with uncontrolled hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, gastrointestinal, or neurological disease are excluded. Participants beginning a new medication or dose changed within the previous 3 months will also be excluded
8. Participants with diagnosed hypertension and/or diabetes
9. Current smoker of cigarette or tobacco, or quit smoking less than 6 months ago, or consume any other inhalable substance, legal or otherwise
10. History of hospitalization or in-patient or out-patient treatment for alcohol or drug dependence or addiction within the 12 months prior to screening. Also, current problem of drug or alcohol abuse which, in the opinion of the investigator, might interfere with participation
11. History of hospitalization or in-patient treatment for depression or any related condition within the past five years. However, use of anti-anxiety/depressants is accepted as long as the dose has been consistent for a minimum of 3 months
12. Chronic or relapsing inflammatory and/or allergic skin conditions such as atopic dermatitis, rosacea, psoriasis and alike including telangiectasias ("spider veins")
13. Current diagnosis of adult acne or currently on treatment for adult acne
14. Participants using tanning salons or tanning products for face in the last 3 months from screening or planning to use them during the study
15. Participants who plan to undergo invasive facial procedures (injections, chemical peeling, etc.) during the study or have undergone these procedures within 1 month prior to baseline
16. Participants with auto-immune skin diseases (e.g., scleroderma, psoriasis, lupus, epidermolysis bullosa, bullous pemphigoid, temporal arteritis)
17. Participant with any current or recent use of medications, treatments, or supplements prohibited/restricted in the protocol
18. Receipt or use of test product(s) in another research study within 30 days prior to baseline visit
19. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant or the quality of the study data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
To assess the effect of Astaxanthin on oxidative stress within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in plasma/serum total antioxidant capacity

SECONDARY OUTCOMES:
To assess the effect of the Astaxanthin on inflammation within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in c-reactive protein
To assess the effect of the Astaxanthin on inflammation within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in tumour necrosis factor alpha
To assess the effect of the Astaxanthin on inflammation within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in Interleukin-6 and Interleukin-10
To assess the effect of the Astaxanthin on lipid levels within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in total cholesterol, high density lipoprotein, low density lipoprotein, and triglycerides
To assess the effect of the Astaxanthin on blood flow within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in blood flow rate and velocity of the brachial artery (volar forearm), as assessed by laser doppler
To assess the effect of the Astaxanthin on facial skin hydration within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in Trans epidermal water loss measurement on the face
To assess the effect of the Astaxanthin on visual skin markers (wrinkles, pores, visible spots, tonality (complexion - even skin tone), pigmentation, roughness (texture), UV porphyrins) after 12 weeks within the group and compared to placebo | 12 weeks
  Change from baseline in Vaestro skin image analysis values from VISIA images
To assess the effect of the Astaxanthin on measures of longevity within the group and compared to placebo | 12 weeks
  Change from baseline in telomere length
To assess the effect of the Astaxanthin on participant reported mood states within the group and compared to placebo | 4 and 12 weeks
  Change from baseline in mood states. Mood states will be measured by Profile of Mood States (POMS) questionnaire that measures feelings description on a 5-point Likert scale ranging from 0 "not at all" to 4 "extremely"
To assess the effect of the Astaxanthin on participant reported facial skin satisfaction within the group and compared to placebo | 4 and 12 weeks
  Self-perceived facial skin satisfaction will be assessed by a self reported short skin questionnaire completed by participants. The questionnaire measures responses on a 5-point Likert scale ranging from "strongly agree" to "strongly disagree"
To assess the safety and tolerability of the Astaxanthin in healthy participants | 12 weeks
  Measurement of Vitals (systolic blood pressure and diastolic blood pressure)
To assess the safety and tolerability of the Astaxanthin in healthy participants | Over 12 weeks
  Collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shoná Burkes-Henderson, PhD, Principal Investigator — SGS Stephens, Inc
Locations (1):
- SGS Stephens, Inc, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No